CLINICAL TRIAL: NCT00664846
Title: Standard Medical Management in Secondary Prevention of Ischemic Stroke in China.
Acronym: SMART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Liying Cui, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2006BAI01A10-1
Record Dates: First submitted 2008-04-12; First posted 2008-04-23 (Estimated); Last update posted 2011-04-11 (Estimated); Status verified 2011-02

CONDITIONS: Stroke
Keywords: Stroke; Prevention Therapy
MeSH Terms: conditions — Stroke | interventions — Aspirin; Clopidogrel; Atorvastatin; Simvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Aspirin / Clopidogrel, Atorvastatin / Simvastatin
- 2 (Active Comparator)
  Interventions: Drug: Asprin / Clopidogrel, Atorvastatin / Simvastatin

INTERVENTIONS:
Drug: Aspirin / Clopidogrel, Atorvastatin / Simvastatin — Standard Medical Management,including antiplatelet agents(Aspirin 75~150mg/day or Clopidogrel 75mg/day),statins(Atorvastatin 20mg/day or Simvastatin 20mg/day),risk factor lowering agents (antihypertension agents:Amlodipine 5mg/day or Benazepril 10mg/day or Valsartan 80mg/day or Nifedipine 30mg/day or Indapamide 2.5mg/day,antidiabetic agents: Metformin 0.5 tid or Glipizide 5mg tid or Acarbose 50mg tid )if necessary,interactive education program (Online medical education program, health behavior guide) .
  Arms: 1
Drug: Asprin / Clopidogrel, Atorvastatin / Simvastatin — Antiplatelet agents(Aspirin 75~150mg/day or Clopidogrel 75mg/day),statins(Atorvastatin 20mg/day or Simvastatin 20mg/day),risk factor lowering agents (antihypertension agents:Amlodipine 5mg/day or Benazepril 10mg/day or Valsartan 80mg/day or Nifedipine 30mg/day or Indapamide 2.5mg/day,antidiabetic agents: Metformin 0.5 tid or Glipizide 5mg tid or Acarbose 50mg tid )if necessary
  Arms: 2

SUMMARY:
The purposes of the study are to analyse the cross-section data of secondary stroke prevention in China and to carry out a standard medical management including medicine and interactive education program,and to evaluate the efficacy and safety of the standard medical management in secondary stroke prevention.

ELIGIBILITY:
Inclusion Criteria:

1. Ischemic cerebral infarction or TIA within 30 days.
2. Aged above 18 years old.
3. Hospitalized.
4. Cranial CT or MRI scan exclude intracranial hemorrhagic diseases
5. Stable clinical and neurological conditions.
6. A Modified Rankin score less than 4 at enrollment
7. Informed consent is obtained.

Exclusion Criteria:

Patients will be excluded from entry if any of the criteria listed below are met

1. Documented stroke caused by conditions other than atherosclerosis, ie, surgical or vascular intervention procedure.
2. Severe co-morbid or unstable medical condition, ie, heart failure, respiratory failure and renal failure, severe liver dysfunction, malignancy with likelihood of death within the next 2 years
3. Significant memory or behavioural disorder, ie, Alzheimer disease, etc, daily care needed.
4. A Modified Rankin score is more than 4
5. Concurrent participation in another clinical trial
6. Pregnant
7. Unable to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4000 (Estimated)
Dates: Start 2008-04; Primary Completion 2010-12 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Success Rate of standard medical management | 1 year after enrolled

SECONDARY OUTCOMES:
Ischemic stroke | 1 year after enrolled
Non-fatal acute coronary syndrome | 1 year after enrolled
Transient Ischemic Attack | 1 year after enrolled
Hemorrhagic Stroke | 1 year after enrolled
All-cause Death | 1 year after enrolled

CONTACTS AND LOCATIONS:
Overall Officials: Liying Cui, Principal Investigator — Peking Union Medical College Hospital
Locations (46):
- China (46):
  - Peking Union Medical College Hosptial, Beijing, Beijing Municipality
  - China Pla General Hospital, Beijing, Beijing Municipality
  - Beijing Daxing District Hospital, Beijing, Beijing Municipality
  - Beijing Ji Shui Tan Hospital,the 4Th Medical College of Peking University, Beijing, Beijing Municipality
  - Beijing Shijitan Hospital, Beijing, Beijing Municipality
  - Beijing Tiantan Hospital, Beijing, Beijing Municipality
  - China Rehabilition Research Center, Beijing, Beijing Municipality
  - General Hospital of Navy, Beijing, Beijing Municipality
  - Luhe Hospital of Tongzhou Distict Beijing, Beijing, Beijing Municipality
  - No 263 Hospital of Pla, Beijing, Beijing Municipality
  - No 309 Hospital of Pla, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Pinggu County Hospital Beijing, Beijing, Beijing Municipality
  - Xuanwu Hospital Capital Medical University, Beijing, Beijing Municipality
  - Daping Hospital, Chongqing, Chongqing Municipality
  - Southwest Hospital, Chongqing, Chongqing Municipality
  - Guangzhou First Municipal People'S Hospital, Guangzhou, Guangdong
  - The First Affiliated Hospital,Sun Yat-Sen Unversity, Guangzhou, Guangdong
  - The First Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The Third Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Yutian County Hospital, Yutian, Hebei
  - Hebei North University, Zhangjiakou, Hebei
  - The First Hospital of Harbin Medical University, Harbin, Helongjiang
  - The Second Hospital of Harbin Medical University, Harbin, Helongjiang
  - Henan Provincial People'S Hospital, Zhengzhou, Henan
  - The Zhongnan Hospital of Wuhan University, Wuhan, Hubei
  - Xiangya Hospital of Centre-South University, Changsha, Hunan
  - Inner Mongolia Baotou City Central Hospital, Baotou, Inner Mongolia
  - The Appurtenant Hospital of Chifeng University, Chifeng, Inner Mongolia
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Nanjing General Hospital of Nanjing Military Command, Nanjing, Jiangsu
  - The Affiliated Drumtower Hospital of Nanjing University Medical School, Nanjing, Jiangsu
  - Jilin University, Changchun, Jilin
  - The Third People'S Hospital of Dalian, Dalian, Liaoning
  - The First Affiliated Hospital of China Medical Sciences University, Shenyang, Liaoning
  - Qinghai Provincial People'S Hospital, Xining, Qinghai
  - Qilu Hospital of Shangdong University, Jinan, Shandong
  - The Second Hospitalof Shangdong University, Jinan, Shandong
  - Huashan Hospital Fudan University, Shanghai, Shanghai Municipality
  - Shanghai Changzheng Hospital, Shanghai, Shanghai Municipality
  - West China Center of Medical Sciences, Chengdu, Sichuan
  - The General Hospital Under Tianjin Medical Sciences University, Tianjin, Tianjin Municipality
  - Tianjin Third Central Hospital, Tianjin, Tianjin Municipality
  - First Affiliated Hospital of Xinjiang Medical University, Uramuqi, Xinjiang Uygur Autonomous Region
  - The First Affiliated Hospital of College of Medicine, Zhejiang University, Hangzhou, Zhejiang

REFERENCES:
- [Derived] Cao Y, Zhang M, Zhou L, Yao M, Peng B, Zhu Y, Ni J, Cui L. Consecutive Slides on Axial View Is More Effective Than Transversal Diameter to Differentiate Mechanisms of Single Subcortical Infarctions in the Lenticulostriate Artery Territory. Front Neurol. 2019 Apr 9;10:336. doi: 10.3389/fneur.2019.00336. eCollection 2019. PMID 31024430
- [Derived] Yao M, Ni J, Zhou L, Peng B, Zhu Y, Cui L; SMART investigators. Elevated Fasting Blood Glucose Is Predictive of Poor Outcome in Non-Diabetic Stroke Patients: A Sub-Group Analysis of SMART. PLoS One. 2016 Aug 5;11(8):e0160674. doi: 10.1371/journal.pone.0160674. eCollection 2016. PMID 27494527
- [Derived] Ni J, Yao M, Zhou L, Zhu Y, Peng B, Cui L; SMART Investigators. A guideline-based program may improve the outcome of stroke among illiterate patients. Int J Stroke. 2016 Apr;11(3):332-7. doi: 10.1177/1747493015626151. Epub 2016 Jan 18. PMID 26780948
- [Derived] Peng B, Ni J, Anderson CS, Zhu Y, Wang Y, Pu C, Wu J, Wang J, Zhou L, Yao M, He J, Shan G, Gao S, Xu W, Cui L; SMART Investigators. Implementation of a structured guideline-based program for the secondary prevention of ischemic stroke in China. Stroke. 2014 Feb;45(2):515-9. doi: 10.1161/STROKEAHA.113.001424. Epub 2014 Jan 2. PMID 24385269
- [Derived] Peng B, Zhu Y, Cui L, Ni J, Xu W, Zhou L, Yao M, Chen L, Wang J, Wang Y, Pu C; SMART Study Group. Standard medical management in secondary prevention of ischemic stroke in China (SMART). Int J Stroke. 2011 Oct;6(5):461-5. doi: 10.1111/j.1747-4949.2011.00648.x. PMID 21951412